CLINICAL TRIAL: NCT01497600
Title: A Randomised, Double-blind, Six-period, Cross-over, Dose-response Trial Investigating the Pharmacodynamics and Pharmacokinetics of Single Doses of Insulin Detemir and NPH Insulin in Subjects of Blacks or African American, Whites of Hispanic or Latino Origin and Whites Not of Hispanic or Latino Origin With Type 2 Diabetes
Brief Title: Pharmacokinetics of Insulin Detemir in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN304-1439
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin detemir (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin NPH
- insulin NPH (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin NPH

INTERVENTIONS:
Drug: insulin detemir — Each subject will be randomly allocated to three doses: 0.3, 0.6, and 1.2 U/kg. Administrated subcutaneously (s.c., under the skin)
Drug: insulin NPH — Each subject will be randomly allocated to three doses: 0.3, 0.6, and 1.2 U/kg. Administrated subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to evaluate the the dose-response of insulin detemir and insulin NPH in subjects with type 2 diabetes of various race and ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Insulin treatment with any insulin preparation/regimen for at least three months with or without combination with below or equal to 2 oral antidiabetic agents (OADs)
* Duration of diabetes at least 12 months
* Body Mass Index (BMI) below 33 kg/m^2
* HbA1c maximum 10 % based on analysis from the central laboratory

Exclusion Criteria:

* Current treatment with insulin above 1.2 U/kg/day
* Current treatment with drugs known to interfere with glucose metabolism other than OADs such as systemic corticosteroids, non-selective beta-blockers, and monoamino oxidase (MAO) inhibitors
* Blood donation of more than 500 mL within the last three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve

SECONDARY OUTCOMES:
Maximum glucose infusion rate
Time to maximum glucose infusion rate.
Area under the serum insulin curve
Maximum serum insulin concentration
Time to maximum insulin concentration
Terminal rate constant of insulin
Terminal half-life of insulin
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Chula Vista, California, United States

REFERENCES:
- [Result] Hompesch M, Troupin B, Heise T, Elbroend B, Endahl L, Haahr H, Heinemann L. Time-action profile of insulin detemir and NPH insulin in patients with type 2 diabetes from different ethnic groups. Diabetes Obes Metab. 2006 Sep;8(5):568-73. doi: 10.1111/j.1463-1326.2006.00643.x. PMID 16918592
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com